CLINICAL TRIAL: NCT05474612
Title: Comparison of Kinesiology Taping and Instrument Assisted Soft Tissue Mobilization in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/01218
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Headache; Cervical Pain
Keywords: Cervicogenic Headache; Instrument Assisted Soft Tissue Mobilization; Kinesiology taping; Cervical range of motion; Neck disability index; Numeric pain rating scale
MeSH Terms: conditions — Headache; Neck Pain; Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: 36 participants were recruited in study and divided into two groups. Group A is given intervention with kinesiology taping and group B is given Instrument Assisted Soft Tissue Mobilization treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiology taping with conventional therapy (Experimental): Patients in group A is treated with conventional treatment (include stretching exercises of SCM, Scaleni and upper fibers of trapezius followed by strengthening (isometrics) of Neck flexors (SCM, rectus capitis, anterior and longus capitis) and then with kinesiology taping.
  Two pieces of the tape cutted in a Y-shape. Applied on deep cervical extensors and upper fibers of trapezius.
  Interventions: Other: kinesiology taping with conventional therapy
- Instrument Assisted Soft Tissue Mobilization with Conventional therapy (Active Comparator): Patients in group B is treated with conventional treatment (stretching exercises of SCM, Scaleni and upper fibers of trapezius followed by strengthening (isometrics) of Neck flexors (SCM, rectus capitis, anterior and longus capitis) and then with Instrument Assisted soft tissue mobilization technique.
  IASTM using tools over the length of targeted muscles (SCM, descending fiber of trapezius, suboccipitalis muscles) in a multidirectional stroking fashion applied to the skin at 30°- 60° for 5 minutes.
  Interventions: Other: Instrument assisted soft tissue mobilization with conventional therapy

INTERVENTIONS:
Other: kinesiology taping with conventional therapy — Two pieces of the tape cutted in a Y-shape. Applied on deep cervical extensors and upper fibers of trapezius. Length of the tape may vary from person to person. Patient is instructed to keep the tape for at-least 2 days.
  Arms: kinesiology taping with conventional therapy
Other: Instrument assisted soft tissue mobilization with conventional therapy — IASTM using tools over the length of targeted muscles (SCM, descending fiber of trapezius, suboccipitalis muscles) in a multidirectional stroking fashion applied to the skin at 30°- 60° for 5 minutes. Participants are in a comfortable position during treatment.
  Arms: Instrument Assisted Soft Tissue Mobilization with Conventional therapy

SUMMARY:
To compare the effects of kinesiology taping and Instrument Assisted Soft Tissue Mobilization in cervicogenic headache

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) is a clinical syndrome characterized by primarily unilateral pain that originates in the neck, typically provoked by neck movement or pressure over tender points in the neck, with reduced range of movement of the cervical spine . It is characterized by unilateral headache with signs and symptoms of neck involvement, such as, pain by movement, by external pressure over the upper cervical, and/or sustained awkward head positions . Functional impairments (diminished strength and endurance) in the cervical muscles and poorer muscle control of the deep cervical flexors have been shown in patients with cervicogenic headache . The International Headache Society (IHS) has declared CGH as a secondary type of headache.The main cause of CGH is dysfunction in the upper cervical spine, and the mechanism of headache involves nociceptive structures such as the disks, upper cervical spinal nerves, facet joints, ganglia, muscles, and ligaments , pain most commonly arises from the second and third cervical spine (C2/3) facet joints, followed by C5/6 facet joints This sign and symptoms are described as the pain being unilateral or bilateral, affecting the head or face but has most commonly affected the occipital region, frontal region, or retro-orbital region, commonly associated with suboccipital neck pain, but can also be associated with ipsilateral arm discomfort. Other symptoms associated with CGH include dizziness, nausea, lightheadedness, inability to concentrate, retro-ocular pain, and visual disturbances.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed cervicogenic headache patients.

* Headache with neck stiffness and pain
* Positive flexion rotation test with restriction 6-10 degree.
* Unilateral headache with referred pattern
* Age between 30-44 years
* Both males and females

Exclusion Criteria:

* Head and neck surgery
* Congenital deformity
* Erosive bone diseases
* Obese
* Disc pathologies
* Malignancy and infection of neck region
* Osteoarthritis
* Rheumatoid arthritis
* Dislocation of vertebraes

Ages: 30 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4th week
  Changes from baseline Numeric pain Rating Scale is used to objectively assess musculoskeletal pain as marked by the patient. It is a 10 point scale from 0 to 10. 0 depicts no pain at all and 10 shows worst pain ever felt. It is measured at baseline and after 4 weeks of the intervention

SECONDARY OUTCOMES:
Neck disability index | 4th week
  Changes from baseline NDI is the most widely used instrument for assessing self-rated disability in patients with neck pain. The NDI is a self-report questionnaire with 10-items. The response to each item is rated on a 6-point scale from 0 (no disability) to 5 (complete disability). The numeric responses for each item are summed for a total score ranging between 0 and 50. Most of the subjects did not know how to drive so their total score is taken from 45. The questionnaire is filled by the subjects at basline and after 4 weeks of the intervention

OTHER OUTCOMES:
inclinometer | 4th week
  Changes from baseline Bubble inclinometers are portable, lightweight, inexpensive and require training. With the movement of neck the ink in the inclinometer moves and the level of ink gives the measure of the range of motion. For flexion, extension and lateral flexion of cervical Range of motion in sitting position and inclinometer is positioned at the top of head in sagittal plane. For rotations the subject is in supine position and inclinometer is placed over the forehead. Cervical ranges of motions are measured at baseline and then after 4 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan